CLINICAL TRIAL: NCT02646059
Title: The Effective Ways of Recruiting Lapsed Blood Donors: a Stratified Randomized Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Principal Investigator, OUYANG Jian, Doctor, Guangzhou Blood Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GuangzhouBC1
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Blood Donor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Text group (Experimental): Text messages containing reminds of blood donation information would be sent to donors in this group.
  Interventions: Other: Text message
- Telephone group (Experimental): Investigators would give telephone calls to the donors in this group, ask the reasons why they stopped donating blood.
  Interventions: Other: Telephone
- Control group (No Intervention): No intervention will be giving to this group.

INTERVENTIONS:
Other: Text message — Text messages would be sent via the messaging platform of Guangzhou Blood Center. The feedback of sending status (received, failed to receive, or unknown) would be marked on every number. Four to six months follow-up, blood donation rate would be checked.
  Arms: Text group
Other: Telephone — Status (response, no answer, line issue, wrong number or refused to be interviewed) of every donor in this groups would be marked. Four to six months follow-up, blood donation rate would be checked.
  Arms: Telephone group

SUMMARY:
Blood donor recruitment is an important issue in every country, since the blood supply pressure become more and more intense. Donor retention is even more important, because it is easier to recruit an old customers than a new one. Therefore, figuring the most effective ways of recruiting lapsed blood donors and understanding the reasons of not donating blood again is critical and vital for the development of blood donation.

ELIGIBILITY:
Inclusion Criteria:

* Donated blood at least once between 2009 to 2013, and the blood test result is qualified.

Exclusion Criteria:

* Having donated again before intervened.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1188 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Blood donation rate | four to six months
  Number of blood donors donate blood again divided by the number of participants in every group after intervened.

SECONDARY OUTCOMES:
Reasons of not donating again | 1 months
  The reasons of not donating again in the telephone group.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China